CLINICAL TRIAL: NCT04891770
Title: A Phase 2a, Open-Label Study to Evaluate the Safety and Efficacy of Selgantolimod (SLGN)-Containing Combination Therapies for the Treatment of Chronic Hepatitis B (CHB)
Brief Title: Study to Evaluate the Safety and Efficacy of Selgantolimod (SLGN)-Containing Combination Therapies for the Treatment of Chronic Hepatitis B (CHB)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Collaborators: Vir Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-465-4439; 2021-000672-11 (EudraCT Number)
Record Dates: First submitted 2021-05-14; First posted 2021-05-18 (Actual); Results first posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — tenofovir alafenamide; Nivolumab; selgantolimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Cohort 1: TAF + VIR-2218 + SLGN + Nivolumab (Experimental): Nucleos(t)ide(s) (NUC)-suppressed participants with chronic hepatitis B (CHB) will receive tenofovir alafenamide (TAF) 25 mg orally once daily (QD) for 36 weeks and VIR-2218 200 mg subcutaneously (SC) once every 4 weeks (Q4W) for 24 weeks. From Week 12 onwards, participants will receive selgantolimod (SLGN) 3 mg orally once a week (QW) for 24 weeks and nivolumab 0.3 mg/kg intravenously (IV) Q4W for up to 24 weeks (only up to protocol amendment 2, nivolumab was no longer administered post implementation of protocol amendment 2). Participants who are on TAF treatment will continue TAF treatment over the duration of study follow-up. Participants will be followed up for 48 weeks post treatment.
  Interventions: Drug: Tenofovir Alafenamide; Drug: VIR-2218; Drug: Nivolumab; Drug: Selgantolimod
- Cohort 2 Group A: VIR-2218 + SLGN + Nivolumab (Experimental): Viremic participants with CHB will receive VIR-2218, 200 mg SC Q4W for 24 weeks. From Week 12 onwards, participants will receive SLGN 3 mg orally QW for 24 weeks and nivolumab 0.3 mg/kg IV Q4W for up to 24 weeks (only up to protocol amendment 2, nivolumab was no longer administered post implementation of protocol amendment 2). Participants who meet the criteria to initiate NUC treatment will receive TAF 25, mg orally, QD during the study. Participants will be followed up for 48 weeks post treatment.
  Interventions: Drug: Tenofovir Alafenamide; Drug: VIR-2218; Drug: Nivolumab; Drug: Selgantolimod
- Cohort 2 Group B: SLGN + Nivolumab (Experimental): Viremic participants with CHB will receive SLGN 3 mg orally QW for 24 weeks and nivolumab 0.3 mg/kg IV Q4W for up to 24 weeks. .
  Viremic participants who meet the criteria to initiate NUC treatment will receive TAF 25 mg orally QD during the study. Participants will be followed up for 48 weeks post treatment.
  All treatments were administered up to protocol amendment 2 and after the implementation of protocol amendment 2, the treatments were discontinued for Cohort 2 Group B based on Sponsor decision.
  Interventions: Drug: Tenofovir Alafenamide; Drug: Nivolumab; Drug: Selgantolimod

INTERVENTIONS:
Drug: Tenofovir Alafenamide — Administered as film-coated oral tablets
  Other Names: TAF; Vemlidy®; GS-7340
Drug: VIR-2218 — Administered as a sub-cutaneous (SC) injection
  Arms: Cohort 1: TAF + VIR-2218 + SLGN + Nivolumab; Cohort 2 Group A: VIR-2218 + SLGN + Nivolumab
Drug: Nivolumab — Administered intravenously
  Other Names: Opdivo®
Drug: Selgantolimod — Administered as film-coated oral tablets
  Other Names: SLGN; GS-9688

SUMMARY:
The primary objectives of this study are to evaluate the safety and tolerability of study treatment(s) (selgantolimod-containing combination therapies) and to evaluate the efficacy of study treatment(s) as measured by the proportion of participants who achieve functional cure, defined as hepatitis B surface antigen (HBsAg) loss and hepatitis B virus (HBV)deoxyribonucleic acid (DNA) < lower limit of quantitation (LLOQ) at Follow-up (FU) Week 24 in participants with chronic hepatitis B (CHB).

ELIGIBILITY:
Key Inclusion Criteria:

* Willing and able to provide informed consent
* Chronic HBV infection for at least 6 months
* Willing to follow protocol-specified contraception requirement

Key Exclusion Criteria:

* Have extensive fibrosis or cirrhosis in the liver
* Have or had liver cancer (hepatocellular carcinoma)
* Have an autoimmune disease
* Have chronic liver disease other than HBV
* Females who are breastfeeding, pregnant, or who wish to become pregnant during the study

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2021-08-14 (Actual); Primary Completion 2024-01-23 (Actual); Study Completion 2024-07-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (26):
- Australia (2):
  - Liverpool Hospital, Liverpool, New South Wales
  - Royal Melbourne Hospital, Parkville, Victoria
- Denmark (4):
  - Aalborg University Hospital, Aalborg
  - Aarhus University Hospital, Aarhus N
  - Hvidovre Hospital, Hvidovre
  - Odense University Hospital, Odense
- Hong Kong (4):
  - Princess Margaret Hospital (Hong Kong), Hong Kong
  - Queen Mary Hospital, Hong Kong
  - Prince of Wales Hospital, Shatin
  - Alice Ho Miu Ling Nethersole Hospital, Tai Po
- Auckland City Hospital, Grafton, New Zealand
- Singapore (3):
  - National University Hospital, Singapore
  - Changi General Hospital, Singapore
  - Singapore General Hospital, Singapore
- South Korea (7):
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul Saint Mary Hospital, Seoul
  - Chung-Ang University Hospital, Seoul
  - Yonsei University Severance Hospital, Seoul
  - Korea University Guro Hospital, Seoul
- Thailand (4):
  - Thai Red Cross AIDS Research Centre (HIV-NAT), Bangkok
  - Ramathibodi Hospital, Bangkok
  - Siriraj Hospital, Bangkok
  - Chiang Mai University, Maharaj Nakorn Chiang Mai Hospital, Muang
- King's College Hospital NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wong GL, Lim SG, Agarwal K, Avihingsanon A, Lim Y, et al. Results From a Phase 2a, Open-Label Study to Evaluate the Safety and Efficacy of Novel Combination Therapies Containing VIR-2218, Selgantolimod, and Nivolumab for the Treatment of Chronic Hepatitis B. Poster #1380; Presented at The Liver Meeting, American Association for the Study of Liver Diseases; 2024 November 15-19; San Diego, CA.
- [Background] Pan D, Kolhatkar N, Sowah L, Arizpe A, Cloutier D, et al. Immunologic Biomarker Dynamics in Chronic Hepatitis B: Insights From a Phase 2a Open-Label Study on Combination Therapies With Small Interfering RNA, Selgantolimod, and Nivolumab. Poster #1134; Presented at The Liver Meeting, American Association for the Study of Liver Diseases; 2024 November 15-19; San Diego, CA.
- [Background] Gane EJ, Tanwandee T, Yi B, Chew T, Botros I, et al. Immune-Related Adverse Events With Low-Dose Nivolumab in Patients With Chronic Hepatitis B: Experience From 3 Clinical Studies. Poster #1332; Presented at The Liver Meeting, American Association for the Study of Liver Diseases; 2024 November 15-19; San Diego, CA.
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study/?id=GS-US-465-4439

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in Australia, Denmark, Hong Kong, New Zealand, Singapore, South Korea, Thailand, and the United Kingdom.
Pre-assignment Details: 165 participants were screened.
Groups:
- Cohort 1: TAF + VIR-2218 + SLGN + Nivolumab: Nucleos(t)ide(s) (NUC)-suppressed participants with chronic hepatitis B (CHB) received tenofovir alafenamide (TAF) 25 mg orally once daily (QD) for 36 weeks and VIR-2218 200 mg subcutaneously (SC) once every 4 weeks (Q4W) for 24 weeks. From Week 12 onwards, participants also received selgantolimod (SLGN) 3 mg orally once a week (QW) for 24 weeks and nivolumab 0.3 mg/kg intravenously (IV) Q4W for up to 24 weeks (only up to protocol amendment 2, nivolumab was no longer administered post implementation of protocol amendment 2). Participants who were on TAF treatment continued TAF treatment over the duration of study follow-up. Participants were followed up for 48 weeks post treatment.
- Cohort 2 Group A: VIR-2218 + SLGN + Nivolumab: Viremic participants with CHB received VIR-2218, 200 mg SC Q4W for 24 weeks. From Week 12 onwards, participants also received SLGN 3 mg orally QW for 24 weeks and nivolumab 0.3 mg/kg IV Q4W for up to 24 weeks (only up to protocol amendment 2, nivolumab was no longer administered post implementation of protocol amendment 2). Participants who met the criteria to initiate NUC treatment received TAF 25, mg orally, QD during the study. Participants were followed up for 48 weeks post treatment.
- Cohort 2 Group B: SLGN + Nivolumab: Viremic participants with CHB received SLGN 3 mg orally QW for 24 weeks and nivolumab 0.3 mg/kg IV Q4W for up to 24 weeks.
  Viremic participants who met the criteria to initiate NUC treatment received TAF 25 mg orally QD during the study. Participants were followed up for 48 weeks post treatment.
  All treatments were administered up to protocol amendment 2 and after the implementation of protocol amendment 2, the treatments were discontinued for Cohort 2 Group B based on Sponsor decision.
Period: Overall Study
Arm/Group | Cohort 1: TAF + VIR-2218 + SLGN + Nivolumab | Cohort 2 Group A: VIR-2218 + SLGN + Nivolumab | Cohort 2 Group B: SLGN + Nivolumab
Started | 42 | 40 | 21
Completed | 41 | 36 | 20
Not Completed | 1 | 4 | 1
Not completed — Withdrew consent | 1 | 3 | 0
Not completed — Enrolled but never treated | 0 | 0 | 1
Not completed — Investigator's discretion | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all participants who received at least 1 dose of study drug.
Groups:
- Cohort 1: TAF + VIR-2218 + SLGN + Nivolumab: NUC -suppressed participants with CHB received TAF 25 mg orally QD for 36 weeks and VIR-2218 200 mg SC Q4W for 24 weeks. From Week 12 onwards, participants also received SLGN 3 mg orally QW for 24 weeks and nivolumab 0.3 mg/kg IV Q4W for up to 24 weeks (only up to protocol amendment 2, nivolumab was no longer administered post implementation of protocol amendment 2). Participants who were on TAF treatment continued TAF treatment over the duration of study follow-up. Participants were followed up for 48 weeks post treatment.
- Total: Total of all reporting groups
Arm/Group | Cohort 1: TAF + VIR-2218 + SLGN + Nivolumab | Cohort 2 Group A: VIR-2218 + SLGN + Nivolumab | Cohort 2 Group B: SLGN + Nivolumab | Total
Number analyzed (Participants) | 42 | 40 | 20 | 102
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 42 | 40 | 20 | 102
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 48 (8.1) | 42 (7.9) | 44 (7.9) | 45 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 25 | 10 | 51
  Male | 26 | 15 | 10 | 51
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: For Ethnicity, data was not collected for 2 participants in the Cohort 1: TAF + VIR-2218 + SLGN + Nivolumab group and for 1 participant in the Cohort 2 Group A: VIR-2218+ SLGN + Nivolumab group.
  Participants
    number analyzed (Participants) | 40 | 39 | 20 | 99
    Hispanic or Latino | 0 | 0 | 0 | 0
    Not Hispanic or Latino | 40 | 39 | 20 | 99
    Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 41 | 37 | 18 | 96
  Race: Black or African American | 1 | 2 | 0 | 3
  Race: Other or More Than One Race | 0 | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  New Zealand | 2 | 1 | 2 | 5
  South Korea | 6 | 2 | 1 | 9
  Singapore | 2 | 8 | 4 | 14
  Hong Kong | 19 | 10 | 7 | 36
  Denmark | 1 | 1 | 0 | 2
  United Kingdom | 2 | 3 | 0 | 5
  Thailand | 8 | 13 | 5 | 26
  Australia | 2 | 2 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved Functional Cure
Description: Functional cure was defined as hepatitis B surface antigen (HBsAg) loss and hepatitis B virus (HBV) deoxyribonucleic acid (DNA) less than the lower limit of quantitation (LLOQ) at follow-up Week 24. LLOQ for HBV DNA CAP/CTM 2.0 is 20 IU/mL. LLOQ for HBV DNA Cobas 6800 is 10 IU/mL. The HBsAg loss was defined as HBsAg changing from positive at baseline to negative at any postbaseline visit. Percentages were rounded off.
Time Frame: At Follow-up Week 24 (Cohort 1 and Cohort 2A: At Week 60; Cohort 2B: At Week 48)
Population: The Full Analysis Set included all enrolled participants in Cohort 1, or all randomized participants in Cohort 2 who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: TAF + VIR-2218 + SLGN + Nivolumab | Cohort 2 Group A: VIR-2218 + SLGN + Nivolumab | Cohort 2 Group B: SLGN + Nivolumab
Number analyzed (Participants) | 42 | 40 | 20
percentage of participants | 2.4 [0.1 to 12.6] | 2.5 [0.1 to 13.2] | 0.0 [0.0 to 16.8]
Statistical Analysis 1: Comparison: Cohort 2 Group A: VIR-2218 + SLGN + Nivolumab vs Cohort 2 Group B: SLGN + Nivolumab; Test type: Other; percentage difference = 2.5, 95% CI 2-sided [-2.3 to 7.3] — For Cohort 2A versus Cohort 2B, the percentage difference and the corresponding 95% confidence interval was calculated using the stratum-adjusted Mantel-Haenszel method, stratified by HBsAg group (> 3 and ≤ 3 log10 IU/mL)

2. Secondary Outcome: Percentage of Participants With HBsAg Loss With and Without Anti-HBsAg Seroconversion
Description: HBsAg loss was defined as HBsAg changing from positive at baseline to negative at any postbaseline visit. HBsAg seroconversion was defined as HBsAg loss and HBsAb changes from negative/missing at baseline to positive at a postbaseline visit. Percentages were rounded-off.
Time Frame: Up to Follow-up Week 48 (Cohort 1 and Cohort 2A: At Week 84; Cohort 2B: At Week 72)
Population: Participants in the Full Analysis Set were analyzed. In Cohort 2 Group B, participants received study treatment for up to 24 weeks. Thereafter, participants were followed up for 48 weeks. Therefore, data for Weeks 28, 32, and 36 are not reported for this cohort in this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: TAF + VIR-2218 + SLGN + Nivolumab | Cohort 2 Group A: VIR-2218 + SLGN + Nivolumab | Cohort 2 Group B: SLGN + Nivolumab
Number analyzed (Participants) | 42 | 40 | 20
percentage of participants
  HBsAg Loss: Week 4 | 0 | 0 | 0
  HBsAg Loss and Seroconversion: Week 4 | 0 | 0 | 0
  HBsAg Loss: Week 8 | 0 | 0 | 0
  HBsAg Loss and Seroconversion: Week 8 | 0 | 0 | 0
  HBsAg Loss: Week 12 | 2.4 | 0 | 0
  HBsAg Loss and Seroconversion: Week 12 | 0 | 0 | 0
  HBsAg Loss: Week 14 | 2.4 | 0 | 0
  HBsAg Loss and Seroconversion: Week 14 | 0 | 0 | 0
  HBsAg Loss: Week 16 | 0 | 0 | 0
  HBsAg Loss and Seroconversion: Week 16 | 0 | 0 | 0
  HBsAg Loss: Week 20 | 4.8 | 2.5 | 0
  HBsAg Loss and Seroconversion: Week 20 | 0 | 0 | 0
  HBsAg Loss: Week 24 | 4.8 | 0 | 0
  HBsAg Loss and Seroconversion: Week 24 | 0 | 0 | 0
  HBsAg Loss: Week 28: number analyzed (Participants) | 42 | 40 | 0
  HBsAg Loss: Week 28 | 4.8 | 0 |
  HBsAg Loss and Seroconversion: Week 28: number analyzed (Participants) | 42 | 40 | 0
  HBsAg Loss and Seroconversion: Week 28 | 0 | 0 |
  HBsAg Loss: Week 32: number analyzed (Participants) | 42 | 40 | 0
  HBsAg Loss: Week 32 | 4.8 | 0 |
  HBsAg Loss and Seroconversion: Week 32: number analyzed (Participants) | 42 | 40 | 0
  HBsAg Loss and Seroconversion: Week 32 | 0 | 0 |
  HBsAg Loss: Week 36: number analyzed (Participants) | 42 | 40 | 0
  HBsAg Loss: Week 36 | 4.8 | 0 |
  HBsAg Loss and Seroconversion: Week 36: number analyzed (Participants) | 42 | 40 | 0
  HBsAg Loss and Seroconversion: Week 36 | 0 | 0 |
  HBsAg Loss: Follow-up (FU) Week 2 | 4.8 | 0 | 0
  HBsAg Loss and Seroconversion: FU Week 2 | 0 | 0 | 0
  HBsAg Loss: FU Week 4 | 4.8 | 0 | 0
  HBsAg Loss and Seroconversion: FU Week 4 | 0 | 0 | 0
  HBsAg Loss: FU Week 8 | 4.8 | 0 | 0
  HBsAg Loss and Seroconversion: FU Week 8 | 0 | 0 | 0
  HBsAg Loss: FU Week 12 | 7.1 | 0 | 0
  HBsAg Loss and Seroconversion: FU Week 12 | 0 | 0 | 0
  HBsAg Loss: FU Week 24 | 4.8 | 2.5 | 0
  HBsAg Loss and Seroconversion: FU Week 24 | 0 | 0 | 0
  HBsAg Loss: FU Week 36 | 7.1 | 2.5 | 0
  HBsAg Loss and Seroconversion: FU Week 36 | 2.4 | 0 | 0
  HBsAg Loss: FU Week 48 | 7.1 | 2.5 | 0
  HBsAg Loss and Seroconversion: FU Week 48 | 0 | 0 | 0

3. Secondary Outcome: Percentage of Participants With Hepatitis B e Antigen (HBeAg) Loss With and Without Anti-HBeAg Seroconversion in Participants With CHB Who Are HBeAg-Positive at Baseline
Description: HBeAg loss is defined as HBeAg changing from positive at baseline to negative at any postbaseline visit. HBeAg seroconversion was defined as HBeAb test changing from negative or missing at baseline to positive at a postbaseline visit. Percentages were rounded-off.
Time Frame: Up to Follow-up Week 48 (Cohort 1 and Cohort 2A: At Week 84; Cohort 2B: At Week 72)
Population: Participants in the Full Analysis Set with HBeAg positive at Baseline were analyzed. In Cohort 2 Group B, participants received study treatment for up to 24 weeks. Thereafter, participants were followed up for 48 weeks. Therefore, data for Weeks 28, 32, and 36 are not reported for this cohort in this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: TAF + VIR-2218 + SLGN + Nivolumab | Cohort 2 Group A: VIR-2218 + SLGN + Nivolumab | Cohort 2 Group B: SLGN + Nivolumab
Number analyzed (Participants) | 18 | 16 | 6
percentage of participants
  HBeAg Loss: Week 4 | 5.6 | 0 | 0
  HBeAg Loss and Seroconversion: Week 4 | 0 | 0 | 0
  HBeAg Loss: Week 8 | 11.1 | 6.3 | 0
  HBeAg Loss and Seroconversion: Week 8 | 0 | 0 | 0
  HBeAg Loss: Week 12 | 11.1 | 6.3 | 0
  HBeAg Loss and Seroconversion: Week 12 | 0 | 0 | 0
  HBeAg Loss: Week 14 | 11.1 | 6.3 | 0
  HBeAg Loss and Seroconversion: Week 14 | 0 | 0 | 0
  HBeAg Loss: Week 16 | 11.1 | 6.3 | 0
  HBeAg Loss and Seroconversion: Week 16 | 0 | 0 | 0
  HBeAg Loss: Week 20 | 11.1 | 6.3 | 0
  HBeAg Loss and Seroconversion: Week 20 | 0 | 0 | 0
  HBeAg Loss: Week 24 | 16.7 | 6.3 | 0
  HBeAg Loss and Seroconversion: Week 24 | 5.6 | 0 | 0
  HBeAg Loss: Week 28: number analyzed (Participants) | 18 | 16 | 0
  HBeAg Loss: Week 28 | 16.7 | 6.3 |
  HBeAg Loss and Seroconversion: Week 28: number analyzed (Participants) | 18 | 16 | 0
  HBeAg Loss and Seroconversion: Week 28 | 5.6 | 0 |
  HBeAg Loss: Week 32: number analyzed (Participants) | 18 | 16 | 0
  HBeAg Loss: Week 32 | 11.1 | 0 |
  HBeAg Loss and Seroconversion: Week 32: number analyzed (Participants) | 18 | 16 | 0
  HBeAg Loss and Seroconversion: Week 32 | 5.6 | 0 |
  HBeAg Loss: Week 36: number analyzed (Participants) | 18 | 16 | 0
  HBeAg Loss: Week 36 | 11.1 | 0 |
  HBeAg Loss and Seroconversion: Week 36: number analyzed (Participants) | 18 | 16 | 0
  HBeAg Loss and Seroconversion: Week 36 | 5.6 | 0 |
  HBeAg Loss: FU Week 2 | 5.6 | 6.3 | 0
  HBeAg Loss and Seroconversion: FU Week 2 | 0 | 6.3 | 0
  HBeAg Loss: FU Week 4 | 16.7 | 6.3 | 0
  HBeAg Loss and Seroconversion: FU Week 4 | 5.6 | 6.3 | 0
  HBeAg Loss: FU Week 8 | 11.1 | 6.3 | 0
  HBeAg Loss and Seroconversion: FU Week 8 | 0 | 6.3 | 0
  HBeAg Loss: FU Week 12 | 16.7 | 6.3 | 0
  HBeAg Loss and Seroconversion: FU Week 12 | 5.6 | 6.3 | 0
  HBeAg Loss: FU Week 24 | 5.6 | 12.5 | 0
  HBeAg Loss and Seroconversion: FU Week 24 | 0 | 12.5 | 0
  HBeAg Loss: FU Week 36 | 11.1 | 12.5 | 0
  HBeAg Loss and Seroconversion: FU Week 36 | 0 | 6.3 | 0
  HBeAg Loss: FU Week 48 | 16.7 | 12.5 | 0
  HBeAg Loss and Seroconversion: FU Week 48 | 5.6 | 6.3 | 0

4. Secondary Outcome: Percentage of Participants Who Remain Off NUC Treatment During Follow-Up
Description: NUC treatments included for analysis: adefovir dipivoxil, entecavir, telbivudine, tenofovir, tenofovir alafenamide, tenofovir alafenamide fumarate, tenofovir disoproxil fumarate, and lamivudine. Percentages were rounded-off.
Time Frame: Cohort 1 and Cohort 2A: From Week 36 up to Week 84 and for Cohort 2B: From Week 24 up to Week 72
Population: The Follow-Up Analysis Set included all participants who have at least 1 follow-up visit, after completing or premature discontinued from the study drugs.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: TAF + VIR-2218 + SLGN + Nivolumab | Cohort 2 Group A: VIR-2218 + SLGN + Nivolumab | Cohort 2 Group B: SLGN + Nivolumab
Number analyzed (Participants) | 42 | 36 | 20
percentage of participants | 16.7 | 55.6 | 75.0

5. Secondary Outcome: Percentage of Participants Experiencing Hepatitis B Virus (HBV) Virologic Breakthrough During Study Treatments
Description: Virologic breakthrough was defined as confirmed HBV DNA ≥ LLOQ after 2 consecutive HBV DNA < LLOQ in participants who are complying with NUC therapy or confirmed HBV DNA ≥ 1 log10 IU/mL increase from nadir during study treatments. LLOQ for HBV DNA CAP/CTM 2.0 is 20 IU/mL. LLOQ for HBV DNA Cobas 6800 is 10 IU/mL. Percentages were rounded-off.
Time Frame: Up to 36 Weeks
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: TAF + VIR-2218 + SLGN + Nivolumab | Cohort 2 Group A: VIR-2218 + SLGN + Nivolumab | Cohort 2 Group B: SLGN + Nivolumab
Number analyzed (Participants) | 42 | 40 | 20
percentage of participants | 7.1 | 35.0 | 20.0

ADVERSE EVENTS:
Time Frame: All-cause Mortality: Up to 86.4 weeks; Adverse events: Up to 84 weeks
Description: All-cause Mortality: The All Enrolled Analysis Set included all participants in Cohort 1 who received a study participant identification number in the study after screening, or all participants in Cohort 2 who were randomized in the study.
  Adverse events: The Safety Analysis Set includes all participants who received at least 1 dose of study drug.
Groups:
- Cohort 1: TAF + VIR-2218 + SLGN + Nivolumab: NUC -suppressed participants with CHB received TAF 25 mg orally QD for 36 weeks and VIR-2218 200 mg SC Q4W for 24 weeks. From Week 12 onwards, participants also received SLGN 3 mg orally QW for 24 weeks and nivolumab 0.3 mg/kg IV Q4W for up to 24 weeks (only up to protocol amendment 2, nivolumab was no longer administered post implementation of protocol amendment 2). Participants who were on TAF treatment continued TAF treatment over the duration of study follow-up for 48 weeks. Participants were followed up for 48 weeks post treatment.
- Cohort 2 Group A: VIR-2218 + SLGN + Nivolumab: Viremic participants with CHB received VIR-2218, 200 mg SC Q4W for 24 weeks. From Week 12 onwards, participants also received SLGN 3 mg orally QW for 24 weeks and nivolumab 0.3 mg/kg IV Q4W for up to 24 weeks (only up to protocol amendment 2, nivolumab was no longer administered post implementation of protocol amendment 2). Participants who met the criteria to initiate NUC treatment received TAF 25, mg orally, QD, for up to 36 weeks during the study. Participants were followed up for 48 weeks post treatment.
- Cohort 2 Group B: SLGN + Nivolumab: Viremic participants with CHB received SLGN 3 mg orally QW for 24 weeks and nivolumab 0.3 mg/kg IV Q4W for up to 24 weeks. .
  Viremic participants who met the criteria to initiate NUC treatment received TAF 25 mg orally QD for up to 36 weeks during the study. Participants were followed up for 48 weeks post treatment.
  All treatments were administered up to protocol amendment 2 and after the implementation of protocol amendment 2, the treatments were discontinued for Cohort 2 Group B based on Sponsor decision.
Arm/Group | Cohort 1: TAF + VIR-2218 + SLGN + Nivolumab | Cohort 2 Group A: VIR-2218 + SLGN + Nivolumab | Cohort 2 Group B: SLGN + Nivolumab
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/40 | 0/21
Serious Adverse Events (participants affected / at risk) | 2/42 | 5/40 | 3/20
Other Adverse Events (participants affected / at risk) | 34/42 | 37/40 | 19/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: TAF + VIR-2218 + SLGN + Nivolumab (N=42) | Cohort 2 Group A: VIR-2218 + SLGN + Nivolumab (N=40) | Cohort 2 Group B: SLGN + Nivolumab (N=20)
Malaise (General disorders) | 0 | 0 | 1
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 | 1 | 0
Chronic hepatitis B (Infections and infestations) | 0 | 1 | 0
Covid-19 (Infections and infestations) | 1 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1
Adenomyosis (Reproductive system and breast disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: TAF + VIR-2218 + SLGN + Nivolumab (N=42) | Cohort 2 Group A: VIR-2218 + SLGN + Nivolumab (N=40) | Cohort 2 Group B: SLGN + Nivolumab (N=20)
Anaemia (Blood and lymphatic system disorders) | 0 | 3 | 0
Palpitations (Cardiac disorders) | 1 | 2 | 0
Conjunctivitis allergic (Eye disorders) | 0 | 1 | 1
Dry eye (Eye disorders) | 0 | 0 | 1
Eye pain (Eye disorders) | 0 | 0 | 1
Ocular discomfort (Eye disorders) | 0 | 0 | 1
Optic neuropathy (Eye disorders) | 0 | 0 | 1
Pseudopapilloedema (Eye disorders) | 0 | 0 | 1
Vision blurred (Eye disorders) | 0 | 1 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 7 | 3
Dyspepsia (Gastrointestinal disorders) | 3 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1
Lip ulceration (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 16 | 27 | 10
Vomiting (Gastrointestinal disorders) | 8 | 15 | 9
Chills (General disorders) | 7 | 4 | 2
Fatigue (General disorders) | 4 | 7 | 4
Injection site pain (General disorders) | 0 | 6 | 0
Injection site reaction (General disorders) | 0 | 2 | 0
Malaise (General disorders) | 0 | 1 | 2
Pyrexia (General disorders) | 4 | 5 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 3 | 2
Seasonal allergy (Immune system disorders) | 0 | 2 | 0
Anal abscess (Infections and infestations) | 1 | 0 | 1
Body tinea (Infections and infestations) | 0 | 0 | 1
Covid-19 (Infections and infestations) | 16 | 10 | 4
Cystitis (Infections and infestations) | 0 | 0 | 1
Fungal skin infection (Infections and infestations) | 0 | 0 | 1
Hepatitis B (Infections and infestations) | 0 | 2 | 0
Influenza (Infections and infestations) | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Otitis externa (Infections and infestations) | 0 | 0 | 1
Periodontitis (Infections and infestations) | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 2
Vulvovaginal candidiasis (Infections and infestations) | 0 | 0 | 1
Eye injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Synovial rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Alanine aminotransferase abnormal (Investigations) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 2 | 11 | 4
Aspartate aminotransferase increased (Investigations) | 2 | 4 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 1 | 1
Dizziness (Nervous system disorders) | 4 | 6 | 2
Dysgeusia (Nervous system disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 6 | 6 | 4
Insomnia (Psychiatric disorders) | 1 | 2 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 1
Heavy menstrual bleeding (Reproductive system and breast disorders) | 0 | 0 | 1
Menstruation irregular (Reproductive system and breast disorders) | 0 | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 3 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Wisdom teeth removal (Surgical and medical procedures) | 0 | 0 | 1
Hypertension (Vascular disorders) | 3 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2023-04-12): https://cdn.clinicaltrials.gov/large-docs/70/NCT04891770/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-18): https://cdn.clinicaltrials.gov/large-docs/70/NCT04891770/SAP_001.pdf